CLINICAL TRIAL: NCT06560749
Title: Physical Exercise for Cognitive Rehabilitation of Patients With Bipolar Affective Disorder: a Controlled and Randomized Study
Brief Title: Physical Exercise for Cognitive Rehabilitation of Patients With Bipolar Affective Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beny Lafer (Other)
Responsible Party: Sponsor-Investigator, Beny Lafer, Principal INvestigator, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 05440818.0.0000.0068
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The experimental group will be submitted to supervised training sessions, three times per week, for 12 weeks, of aerobics exercises, as well as treatment as usual (TAU)
  Interventions: Other: Physical Exercise
- Control Group (No Intervention): the control group will be submitted exclusively to treatment as usual (TAU)

INTERVENTIONS:
Other: Physical Exercise — Measure the impact of physical exercise in the cognition of pacients diagnosed with Bipolar Disorder
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate the impact of Physical Exercise (PE), as an adjuvant treatment, on the cognition of patients diagnosed with Bipolar Disorder who present cognitive impairments, as well as its impact on quality of life and functionality and its association with physiological variables.

Our specific goals are:

1. Evaluate the effect of PE on the neuropsychological functions of attention, memory, verbal fluency, executive function and processing speed in patients diagnosed with BD who present cognitive impairments in these domains.
2. To evaluate the effect of PE on the quality of life and functionality of patients diagnosed with BD, as well as possible associations with cognitive functions.
3. To evaluate possible correlations between physiological variables, such as cardiorespiratory indices, strength and body composition, and improvements in cognitive functions, quality of life and functionality.

DETAILED DESCRIPTION:
The study aims to assess the impact of structured physical exercise on the cognitive function of bipolar disorder patients presenting deficits, while investigating its association to quality of life and functionality. The study will include 72 euthymic BD patients from the Bipolar Disorder Research Program (PROMAN) at the Institute of Psychiatry of the University of São Paulo Medical School, randomly distributed into two groups: 1) the experimental group will be submitted to supervised training sessions, three times per week, for 12 weeks, including aerobics and strength exercises, as well as treatment as usual (TAU); and 2) the control group will be submitted exclusively to TAU. Cognitive function, depressive and manic symptoms, quality of life and functionality will be assessed at baseline and at follow-uo (week 12), for both groups. Statistical hypothesis testing, assessing the presence of statistically significant differences between groups, pre and post intervention, should be available on the third quarter of 2025.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar disorder (BD) I and II according to DSM-5
* Age: 18 - 55 years old
* Complete primary education
* Euthymic (YMRS < 8 and MADRS < 12)
* Presence of cognitive impairments (COBRA > 14 and SCIP < 75)
* Estimated IQ ≥ 80
* No medication changes in the last month
* Having been without regular PE practice for six months
* Signature of the TCLE

Exclusion Criteria:

* Organic mental disorder
* BMI > 40
* Alcohol or drug abuse in the last 6 months
* Use of benzodiazepines or beta-blockers in the last month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, Week 4, Week 8 and Follow-up (12 weeks)
  Scale used to assess the presence and intensity of depressive symptoms.
Young Mania Rating Scale (YMRS) | Baseline, Week 4, Week 8 and Follow-up (12 weeks)
  Scale used to assess the presence and intensity of manic symptoms.
Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA) | Baseline only
  Screening scale for the presence of cognitive deficits. Suggested cutoff point is 14
Screen for Cognitive Impairment in Psychiatry (SCIP) | Baseline only
  Subjective screening scale for difficulties associated with cognitive impairment. Suggested cutoff point is 70
Stroop Color-Word Test (Spreen and Strauss, 1998) | Baseline and Follow-up (12 weeks)
  Assessing mental flexibility and inhibitory control (attention and executive function)
Verbal Fluency - F.A.S (Spreen and Strauss, 1998) | Baseline and Follow-up (12 weeks)
  Assessing verbal fluency, inhibitory control and the correct use of strategies (executive function)
Trail Making Test (Spreen and Strauss, 1998) | Baseline and Follow-up (12 weeks)
  Assessing alternating attention
Logical Memory I and II (Wechsler, 1997b) | Baseline and Follow-up (12 weeks)
  Assessing verbal memory
List of Words (Wechsler, 1997a) | Baseline and Follow-up (12 weeks)
  Assessing learning capacity and attention
Cardiovascular evaluation | Baseline and Follow-up (12 weeks)
  All patients will undergo an electrocardiogram computerized.
Stress test on the treadmill | Baseline and Follow-up (12 weeks)
  A treadmill stress test will be performed.
Respiratory gas exchange analysis (ergospirometric) | Baseline and Follow-up (12 weeks)
  A computerized gas exchange analysis system will be used (CPX/ULTIMA, Medgraphics®, Saint Paul, MN, USA)
Isokinetic Strength Test | Baseline and Follow-up (12 weeks)
  The isokinetic test will be performed on the lower limbs (extensor and flexor muscles of the knee joints) on the dominant (R) and non-dominant (ND) leg at an angular velocity of 60 s -1 using a computerized isokinetic dynamometer (Biodex®, Inc . USA).
Body composition by bioimpedance | Baseline and Follow-up (12 weeks)
  Body composition measurements will be obtained by the non-invasive indirect bioimpedance method using a scale
Anthropometric measurements (skinfolds) and calculation of body composition | Baseline and Follow-up (12 weeks)
  Body mass (BM) will be measured on a Filizola mechanical scale, with an accuracy of 0.1 kg. Height will be determined using a stadiometer, attached to the scale, with an accuracy of 0.1cm (Gordon et al., 1988). Body composition will be determined using the skinfold thickness technique.
One Repetition Maximum Test (1RM) | Baseline and Follow-up (12 weeks)
  The exercises to be tested are the seated bench press (pectoral muscles), leg-press (quadriceps and glutes), rowing (dorsal muscles), standing knee bending chair (hamstrings), abdominal (rectus and abdominal obliques).
Wechsler Abbreviated Scale of Intelligence (WASI) | Baseline and Follow-up (12 weeks)
  delivers an estimation of a student's general intellectual ability by measuring the verbal, nonverbal, and general cognition of individuals from 6 to 89 years of age.
Digit Span Memory Test | Baseline and Follow-up (12 weeks)
  short test that evaluates a person's memory and cognitive status
Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline and Follow-up (12 weeks)
  Questionnaire measuring cognitive coping strategies
Difficulties in Emotion Regulation Scale (DERS) | Baseline and Follow-up (12 weeks)
  Instrument measuring emotion regulation problems

SECONDARY OUTCOMES:
Functional Assessment Staging Tool (FAST) | Baseline and Follow-up (12 weeks)
  Scale used to assess the patient's global functionality.
The World Health Organization Quality of Life Assessment (WHOQOL) | Baseline and Follow-up (12 weeks)
  Scale used to assess patients quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Beny Lafer, M.D, Ph.D, Principal Investigator — University of Sao Paulo
Locations (1):
- Gabriel Okawa Belizario, São Paulo, São Paulo, Brazil